CLINICAL TRIAL: NCT03176810
Title: Comparison Between Optimal Coherence Tomography Guidance and Angiography Guidance in Percutaneous Coronary Intervention
Acronym: COCOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Takashi Kubo, MD (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor-Investigator, Takashi Kubo, MD, Associate Professor, Wakayama Medical University
Organization: Wakayama Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1856
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Coronary Disease
Keywords: percutaneous coronary intervention; optical coherence tomography
MeSH Terms: conditions — Coronary Disease | interventions — Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided PCI (Active Comparator): PCI is performed by OCT guidance.
  Interventions: Device: OCT
- Angiography-guided PCI (Active Comparator): PCI is performed by angiography guidance alone.
  Interventions: Device: Angiography

INTERVENTIONS:
Device: OCT — OCT is used to guide PCI.
  Arms: OCT-guided PCI
Device: Angiography — Angiography is used to guide PCI.
  Arms: Angiography-guided PCI

SUMMARY:
The present study aims to demonstrate the superiority of optical coherence tomography (OCT)-guided percutaneous coronary intervention (PCI) compared with Angiography-guided PCI.

DETAILED DESCRIPTION:
Comparison between Optimal Coherence tomography guidance and Angiography Guidance in percutaneous coronary intervention (COCOA) is a prospective, multicentre, randomised, open-label, parallel group, active-controlled, superiority trial comparing minimum stent area immediately after optical coherence tomography (OCT)-guided percutaneous coronary intervention (PCI) with those after Angiography-guided PCI with a second generation drug-eluting stent.The primary endpoint of the present study was minimum stent area immediately after PCI. The secondary endpoint was target vessel failure (defined as a composite of cardiac death, target-vessel related myocardial infarction, and ischaemia-driven target vessel revascularisation).

ELIGIBILITY:
Inclusion Criteria:

1. Patients eligible for PCI using drug-eluting stent (DES) to a de novo native coronary artery lesion in stable angina pectoris, unstable angina pectoris or non-ST-segment elevation myocardial infarction (evaluated based on the guideline)
2. Aged 20 years or older at the time of their consent
3. Patients who agree to be enrolled in the trial giving signed written informed consent

Exclusion Criteria:

1) Patients who have showed ST-segment elevation myocardial infarction in previous 3 months 2) Patients with cardiogenic shock 3) Patients with heart failure 4) Patients with 3-vessel disease 5) Patients scheduled to use bare metal stent 6) Patients with renal function disorder (eGFR 30 mL/min/1.73 m2 or less or serum creatinine 1.5 mg/dL or more) 7) Patients undergoing hemodialysis 8) Patients with allergies to aspirin, clopidogrel, prasugrel, heparin, and iodinated contrast agents 9) Patients with hemorrhagic complications such as intracranial hemorrhage and gastrointestinal bleeding 10) Patients scheduled to undergo surgical treatment after PCI within 1 year 11) Patients participating in the clinical study of other medical device or drug and who were considered affecting the primary endpoint of this study by the physician in charge 12) Patients with one or more co-morbidities that shorten life expectancy to less than 12 months or that may interfere with the study process according to this study protocol 13) Patients scheduled to use IVUS in PCI 14) Patients in whom the form of the target disease concerned is applicable to any of the following lesions: (i) Lesion in the previously (within 1 year) treated coronary artery or lesion in the coronary artery with the other lesions requiring revascularization with PCI in the near future (within 1 year) (ii) Lesion in the left main coronary artery (iii) Lesion in the coronary bypass graft (iv) Aorto-ostial lesion in right coronary artery (arising within 3 mm of the origin of a right coronary artery) (v) Lesion of chronic total occlusion (vi) Coronary bifurcation lesion requiring revascularization with 2 stents (vii) Coronary bypass graft lesion (viii) Lesion in coronary artery with diameter of < 2.5mm or >4.00mm (ix) Long lesion (length >40mm) (x) Lesion in coronary artery where we expected difficulty in advancing the OCT catheter (e.g. extremely tortuous artery or severely calcified artery)

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Minimum stent area | Immediately after PCI
  Minimum stent area is measured by OCT

SECONDARY OUTCOMES:
Target vessel failure | 12-month afte PCI
  Target vessel failure is defined as a composite of cardiac death, target-vessel related myocardial infarction, and ischaemia-driven target vessel revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Akaska, MD, Principal Investigator — Wakayama Medical University
Locations (1):
- Department of Cardiovascular Medicine, Wakayama Medical University, Wakayama, Japan

IPD SHARING:
Plan to Share IPD: Undecided